CLINICAL TRIAL: NCT01635686
Title: A Randomized, Double-blind, Single-dosing, Crossover Study to Compare the Safety and Pharmacokinetic Characteristics of DWP422 25 mg With Those of ENBREL 25MG PFS INJ. After Subcutaneous Injection in Healthy Male Volunteers
Brief Title: Comparison the Safety and Pharmacokinetic Characteristics of DWP422 25 mg With Those of ENBREL 25MG PFS INJ. After Subcutaneous Injection in Healthy Male Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double
Other Study IDs: DW_DWP422001
Record Dates: First submitted 2012-07-04; First posted 2012-07-09 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

ARMS (2):
- DWP422 (Experimental)
  Interventions: Drug: DWP422 25mg
- ENBREL (Active Comparator)
  Interventions: Drug: ENBREL 25MG PFS INJ.

INTERVENTIONS:
Drug: DWP422 25mg
  Arms: DWP422
Drug: ENBREL 25MG PFS INJ.
  Arms: ENBREL

SUMMARY:
The purpose of this study was to compare the safety and pharmacokinetic characteristics of DWP422 25 mg with those of ENBREL 25MG PFS INJ. after subcutaneous injection in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males, 20 to 45 years of age the moment of screening
2. Body mass index is between 19.0 and 27.0 kg/m2

Exclusion Criteria:

1. Hypersensitivity response to the experimental and comparator drugs
2. The tuberculosis patient or latent tuberculosis patient

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Etanercept levels in blood

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea